CLINICAL TRIAL: NCT02319044
Title: A Phase II, Randomized, Open-Label, Multi-Center, Global Study of MEDI4736 Monotherapy, Tremelimumab Monotherapy, and MEDI4736 in Combination With Tremelimumab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Phase II Study of MEDI4736, Tremelimumab, and MEDI4736 in Combination w/ Tremelimumab Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4193C00003
Record Dates: First submitted 2014-12-12; First posted 2014-12-18 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Recurrent/Metastatic Squamous Cell Carcinoma of Head & Neck
Keywords: Head and neck cancer; SCCHN
MeSH Terms: conditions — Recurrence; Head and Neck Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI4736 (Experimental): MEDI4736 monotherapy
  Interventions: Drug: MEDI4736
- Tremelimumab (Experimental): Tremelimumab monotherapy
  Interventions: Drug: Tremelimumab
- MEDI4736 + Tremelimumab (Experimental): MEDI4736 + Tremelimumab combination therapy
  Interventions: Drug: MEDI4736 + Tremelimumab

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 monotherapy
  Arms: MEDI4736
Drug: Tremelimumab — Tremelimumab monotherapy
  Arms: Tremelimumab
Drug: MEDI4736 + Tremelimumab — MEDI4736 + Tremelimumab combination therapy
  Arms: MEDI4736 + Tremelimumab

SUMMARY:
The purpose of this study is to determine the efficacy and safety of investigational medical products (MEDI4736 monotherapy, tremelimumab monotherapy, and MEDI4736 + tremelimumab combination therapy) in the treatment of patients with recurrent or metastatic carcinoma of the head and neck who have progressed during or after treatment with a platinum containing regimen for recurrent/metastatic disease.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, global, Phase II study to determine the efficacy and safety of MEDI4736 + tremelimumab combination therapy, MEDI4736 monotherapy and tremelimumab monotherapy in the treatment of patients with recurrent or metastatic PD-L1-negative squamous cell carcinoma of the head and neck (SCCHN) who have progressed during or after treatment with only 1 systemic palliative regimen for recurrent or metastatic disease, that must have contained a platinum agent.

Patients will be randomized in a stratified manner according to prognostic factors, including human papillomavirus (HPV) status and smoking status to achieve a balance between treatments for each of the factors. Patients will be randomized in a 1:1:2 fashion to receive MEDI4736 monotherapy, tremelimumab monotherapy, or MEDI4736 + tremelimumab combination.

All treatments will be administered beginning on Day 0 for 12 months or until confirmed progression of disease; unless, in the Investigator's opinion, the patient continues to receive benefit from the treatment), initiation of alternative cancer therapy, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. Patients with confirmed progression of disease who, in the Investigator's opinion, continue to receive benefit from their assigned investigational product and who meet the criteria for treatment in the setting of progression of disease may continue to receive their assigned investigational product treatment for a maximum of 12 months after consultation with the Sponsor and at the Investigator's discretion. The monotherapy arms (tremelimumab and MEDI4736) should be discontinued if there is confirmed progression of disease following a previous response in target lesions (complete response or partial response).

Tumor assessments will be performed using computed tomography or magnetic resonance imaging. Efficacy for all patients will be assessed by objective tumor assessments every 8 weeks (q8w) for the first 48 weeks (relative to the date of the first infusion) then q12w in patients who have disease control after 12 months until confirmed objective disease progression.

Following completion or discontinuation of treatment, patients will enter a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Written informed consent obtained from the patient/legal representative;
* Histologically confirmed recurrent or metastatic SCCHN; tumor progression or recurrence during or after treatment with only 1 systemic palliative regimen for recurrent or metastatic disease that must have contained a platinum agent; Patients who have only received chemo-radiation with curative intent for treatment of their locally advanced disease or recurrent disease are not eligible. Patients who received concurrent chemo-radiation as part of treatment of their recurrent disease are also not eligible.
* Written consent to provide newly acquired tumor tissue (preferred) or archival tissue for the purpose of establishing PD-L1 status.
* Confirmed PD-L1-negative SCCHN by Ventana SP263;
* WHO/ECOG performance status of 0 or 1;
* At least 1 measurable lesion at baseline;
* No prior exposure to immune-mediated therapy;
* Adequate organ and marrow function; Evidence of post-menopausal status or negative urinary or serum pregnancy test.

Exclusion Criteria:

* Histologically confirmed squamous cell carcinoma of any other primary anatomic location in the head and neck;
* Received more than 1 regimen for recurrent or metastatic disease
* Any concurrent chemotherapy, Investigational Product, biologic, or hormonal therapy for cancer treatment;
* Receipt of any investigational anticancer therapy within 28 days or 5 half-lives;
* Receipt of last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, mAbs, etc) within 21 days prior to the first dose of study treatment;
* Major surgical procedure within 28 days prior to the first dose of Investigational Product;
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criterion;
* Current or prior use of immunosuppressive medication within 14 days before the first dose of their assigned Investigational Product;
* History of allogeneic organ transplantation;
* Active or prior documented autoimmune or inflammatory disorders;
* Uncontrolled intercurrent illness;
* another primary malignancy
* Patients with history of brain metastases, spinal cord compression, or a history of leptomeningeal carcinomatosis;
* History of active primary immunodeficiency;
* Known history of previous tuberculosis;
* Active infection including hepatitis B, hepatitis C or human immunodeficiency virus (HIV);
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of Investigational Product;
* Pregnant or breast-feeding female patients;
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
* Known allergy or hypersensitivity to Investigational Product.
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the IP or interpretation of patient safety or study results

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Wrona, Study Director — Medical Scientist AstraZeneca Magdalena.Wrona@astrazeneca.com; Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital in Toronto, Ontario
Locations (113):
- United States (41):
  - Research Site, Birmingham, Alabama
  - Research Site, Yuma, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Downey, California
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Australia (3):
  - Research Site, Adelaide
  - Research Site, Darlinghurst
  - Research Site, Tweed Heads
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Namur
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Moncton, New Brunswick
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Zlín
- France (16):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Rouen
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Grégoire
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (6):
  - Research Site, Berlin
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, München
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Zalaegerszeg
- Israel (3):
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Tel Litwinsky
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Suwon
- Spain (10):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Zaragoza
- Research Site, Taipei, Taiwan
- United Kingdom (6):
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Siu LL, Even C, Mesia R, Remenar E, Daste A, Delord JP, Krauss J, Saba NF, Nabell L, Ready NE, Brana I, Kotecki N, Zandberg DP, Gilbert J, Mehanna H, Bonomi M, Jarkowski A, Melillo G, Armstrong JM, Wildsmith S, Fayette J. Safety and Efficacy of Durvalumab With or Without Tremelimumab in Patients With PD-L1-Low/Negative Recurrent or Metastatic HNSCC: The Phase 2 CONDOR Randomized Clinical Trial. JAMA Oncol. 2019 Feb 1;5(2):195-203. doi: 10.1001/jamaoncol.2018.4628. PMID 30383184
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3110&filename=Redacted%20CONDOR%20Protocol%2020Sept17.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 127 sites in 15 countries enrolled and screened patients. The study was conducted and managed by PRA, a contract research organization.
Groups:
- MEDI4736 AND TREMELIMUMAB COMBINATION: MEDI4736 (20 mg/kg) + Tremelimumab (1 mg/kg) combination therapy administered via intravenous infusion every 4 weeks for up to 4 months (4 doses), then MEDI4736 (10 mg/kg) as a single agent every 2 weeks to complete 12 months of treatment
- MEDI4736: MEDI4736 (10 mg/kg) monotherapy administered via intravenous infusion every 2 weeks for up to 12 months (up to 26 doses)
- Tremelimumab: Tremelimumab (10 mg/kg) monotherapy administered via intravenous infusion every 4 weeks for 7 doses, then every 12 weeks for 2 additional doses for up to 12 months (up to 9 doses)
Period: Overall Study
Arm/Group | MEDI4736 AND TREMELIMUMAB COMBINATION | MEDI4736 | Tremelimumab
Started | 133 | 67 | 67
Completed | 11 | 7 | 0
Not Completed | 122 | 60 | 67
Not completed — Death, PI/sponsor decision, med history | 0 | 1 | 4
Not completed — Withdrawal by Subject | 3 | 3 | 6
Not completed — Condition under investigation worsened | 100 | 50 | 46
Not completed — Adverse Event | 17 | 2 | 8
Not completed — Study specific discontinuation criteria | 2 | 2 | 1
Not completed — Not treated | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set - all randomized patients
Groups:
- MEDI4736 + Tremelimumab: MEDI4736 (20 mg/kg) + Tremelimumab (1 mg/kg) combination therapy administered via intravenous infusion every 4 weeks for up to 4 months (4 doses), then MEDI4736 (10 mg/kg) as a single agent every 2 weeks to complete 12 months of treatment
- Total: Total of all reporting groups
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 133 | 67 | 67 | 267
Age, Categorical [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 88 | 46 | 42 | 176
    >=65 years | 45 | 21 | 25 | 91
Age, Continuous [Median (Full Range); unit: years] — Population: Full analysis set - all randomized patients
  years | 62 [26 to 81] | 62 [23 to 82] | 61 [42 to 77] | 61 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    Female | 20 | 13 | 14 | 47
    Male | 113 | 54 | 53 | 220
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 4 | 3 | 2 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 6 | 3 | 1 | 10
    White | 115 | 58 | 57 | 230
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 8 | 3 | 7 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    Ethnic group - Hispanic or Latino | 8 | 2 | 5 | 15
    Ethnic group - Not Hispanic or Latino | 119 | 64 | 58 | 241
    Ethnic group - Total | 127 | 66 | 63 | 256
    Asian ethnic group - Asian (not Chinese/Japanese) | 3 | 2 | 1 | 6
    Asian ethnic group - Chinese | 1 | 1 | 1 | 3
    Asian ethnic group - Total | 4 | 3 | 2 | 9
    Unknown or not reported | 2 | 0 | 2 | 4
Negative PD-L1 status [Count of Participants; unit: Participants] — Programmed cell death ligand 1 status identification performed at screening Population: Full analysis set - all randomized patients
  Participants
    PD-L1 negative patients | 133 | 67 | 67 | 267
HPV status [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    Positive | 39 | 18 | 18 | 75
    Negative | 94 | 49 | 49 | 192
Use of nicotine (other than cigarettes) [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    Yes | 1 | 1 | 0 | 2
    No | 132 | 66 | 67 | 265
Smoking/nicotine status by nicotine user [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    Current smoker >10 pack years | 22 | 7 | 6 | 35
    Current smoker <= 10 pack years | 2 | 0 | 1 | 3
    Former smoker >10 pack years | 59 | 35 | 34 | 128
    Former smoker <= 10 pack years | 30 | 16 | 12 | 58
    Never | 20 | 9 | 14 | 43
WHO/ECOG performance status at study entry [Count of Participants; unit: Participants] — Population: Full analysis set - all randomized patients
  Participants
    (0) Normal activity | 40 | 22 | 19 | 81
    (1) Restricted activity | 93 | 45 | 48 | 186

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate at 6 Months
Description: Objective response rate, primary analysis, based on BICR assessments according to RECIST v1.1. The number (%) of patients with a response excludes unconfirmed responses
Time Frame: After 6 months
Population: Evaluable analysis set - all patients who received at least one dose of study treatment, who had a baseline tumor assessment, and had measurable disease
Measure: Number (95% Confidence Interval); unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab
Number analyzed (Participants) | 130 | 65 | 63
% participants | 7.7 [3.75 to 13.69] | 9.2 [3.46 to 19.02] | 1.6 [0.04 to 8.53]

2. Primary Outcome: Objective Response Rate at 12 Months
Description: Objective response rate (per RECIST 1.1 as assessed by blinded independent central review [BICR]) is defined as the number (%) of patients with a confirmed complete response or confirmed partial response and will be based on all treated patients who are PD-L1-positive with measurable disease at baseline per BICR. Response Evaluation Criteria in Solid Tumors [RECIST] 1.1. criteria are: Complete response [CR] = disappearance of all target lesions since baseline; and partial response [PR] = at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab
Number analyzed (Participants) | 129 | 65 | 63
% participants
  Overall | 7.8 [3.78 to 13.79] | 9.2 [3.46 to 19.02] | 1.6 [0.04 to 8.53]
  Current smoking/nicotine status - Total: number analyzed (Participants) | 22 | 7 | 7
  Current smoking/nicotine status - Total | 13.6 [2.91 to 34.91] | 14.3 [0.36 to 57.87] | 14.3 [0.36 to 57.87]
  Current smoking/nicotine status - >10 pack years: number analyzed (Participants) | 20 | 7 | 6
  Current smoking/nicotine status - >10 pack years | 15.0 [3.21 to 37.89] | 14.3 [0.36 to 57.87] | 16.7 [0.42 to 64.12]
  Current smoking/nicotine status - ≤10 pack years: number analyzed (Participants) | 2 | 0 | 1
  Current smoking/nicotine status - ≤10 pack years | 0 [0.00 to 84.19] |  | 0 [0.00 to 97.50]
  Former smoking/nicotine status -Total: number analyzed (Participants) | 88 | 49 | 44
  Former smoking/nicotine status -Total | 6.8 [2.54 to 14.25] | 8.2 [2.27 to 19.60] | 0 [0.00 to 8.04]
  Former smoking/nicotine status - >10 pack years: number analyzed (Participants) | 58 | 33 | 32
  Former smoking/nicotine status - >10 pack years | 5.2 [1.08 to 14.38] | 9.1 [1.92 to 24.33] | 0 [0.00 to 10.89]
  Former smoking/nicotine status - ≤10 pack years: number analyzed (Participants) | 30 | 16 | 12
  Former smoking/nicotine status - ≤10 pack years | 10.0 [2.11 to 26.53] | 6.3 [0.16 to 30.23] | 0 [0.00 to 26.46]
  Smoking/nicotine status - Never: number analyzed (Participants) | 19 | 9 | 12
  Smoking/nicotine status - Never | 5.3 [0.13 to 26.03] | 11.1 [0.28 to 48.25] | 0 [0.00 to 26.46]
  HPV status - Positive: number analyzed (Participants) | 37 | 18 | 18
  HPV status - Positive | 5.4 [0.66 to 18.19] | 16.7 [3.58 to 41.42] | 0 [0.00 to 18.53]
  HPV status - Negative: number analyzed (Participants) | 92 | 47 | 45
  HPV status - Negative | 8.7 [3.83 to 16.42] | 6.4 [1.34 to 17.54] | 2.2 [0.06 to 11.77]

3. Secondary Outcome: Best Objective Response
Description: The best response a patient has had during their time in the study
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number; unit: % participants
Groups:
- Total: Total across all treatment groups
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 129 | 65 | 63 | 257
% participants
  Response - Total | 7.8 | 9.2 | 1.6 | 6.6
  Response - Complete response (CR) | 0 | 0 | 0 | 0
  Response - Partial response (PR) | 7.8 | 9.2 | 1.6 | 6.6
  Non-response (NR) - Total | 92.2 | 90.8 | 98.4 | 93.4
  NR - Stable disease (SD) >=6 months (24 weeks) | 5.4 | 6.2 | 0 | 4.3
  NR - Unconfirmed complete or partial response (PR) | 1.6 | 0 | 0 | 0.8
  NR - Stable disease | 3.9 | 6.2 | 0 | 3.5
  NR - Progression | 64.3 | 64.6 | 69.8 | 65.8
  NR - Progression-RECIST 1.1 progression | 45.7 | 46.2 | 54.0 | 47.9
  NR - Progression-Death | 18.6 | 18.5 | 15.9 | 17.9
  NR - Not evaluable-Total | 22.5 | 20.0 | 28.6 | 23.3
  NR - Not evaluable-SD <6 months (24 weeks) | 20.2 | 16.9 | 19.0 | 19.1
  NR - Not evaluable-Incomplete post baseline tests | 2.3 | 3.1 | 9.5 | 4.3

4. Secondary Outcome: Duration of Response - Participants Remaining in Response
Description: Participants remaining in response - based on BICR assessments according to RECIST v1.1. An ongoing response was defined as a patient who had documented objective response and was still alive and progression-free at the time of the data cut-off.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 10 | 6 | 1 | 17
% participants
  Percentage remaining in response-3 months | 90.0 | 100 | 100 | 94.1
  Percentage remaining in response-6 months | 70.0 | 66.7 | 100 | 70.6
  Percentage remaining in response-9 months | 58.3 | 66.7 | NA — No participants in this category | 64.2
  Percentage remaining in response-12 months | 46.7 | NA — No participants in this category | NA — No participants in this category | 53.5
  Percentage of ongoing response | 50.0 | 66.7 | 100 | 58.8

5. Secondary Outcome: Time to Response
Description: Time to response in patients with objective response based on BICR assessments according to RECIST 1.1
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 10 | 6 | 1 | 17
% participants
  Number of responders | 100 | 100 | 100 | 100
  Week 8, where response is first observed | 10.0 | 0 | 0 | 5.9
  Week 9, where response is first observed | 50.0 | 16.7 | 100 | 41.2
  Week 16, where response is first observed | 10.0 | 16.7 | 0 | 11.8
  Week 17, where response is first observed | 10.0 | 16.7 | 0 | 11.8
  Week 20, where response is first observed | 0 | 16.7 | 0 | 5.9
  Week 24, where response is first observed | 10.0 | 16.7 | 0 | 11.8
  Week 25, where response is first observed | 10.0 | 16.7 | 0 | 11.8

6. Secondary Outcome: Time to Onset of Response From First Dose
Description: Time to onset of response in patients with objective response based on BICR assessments according to RECIST 1.1
Time Frame: After 12 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 10 | 6 | 1 | 17
Months | 2.0 [2 to 6] | 4.1 [2 to 6] | 1.8 [1.8 to 2] | 3.5 [2 to 6]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) at 6 months based on BICR assessments according to RECIST v1.1. DCR at 6 months was evaluated using 2 different approaches to the length of stable disease (SD). -Method 1: Patients who had a best objective response of complete response (CR) or partial response (PR) within 24 weeks or had demonstrated SD for a minimum interval of 24 weeks following randomization. -Method 2: Patients who had a best objective response of CR or PR in the first 24 weeks or who had demonstrated SD for a minimum interval of 16 weeks following randomization.
Time Frame: After 6 months
Population: as for outcome 1
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 129 | 65 | 63 | 257
% participants
  METHOD 1: Disease control (DC) at 6 months | 13.2 | 21.5 | 1.6 | 12.5
  METHOD 1: No DC at 6 months | 86.8 | 78.5 | 98.4 | 87.5
  METHOD 1: No DC at 6 months-Not evaluable/missing | 20.2 | 20.0 | 22.2 | 20.6
  METHOD 2: DC at 6 months | 20.2 | 26.2 | 9.5 | 19.1
  METHOD 2: No DC at 6 months | 79.8 | 73.8 | 90.5 | 80.9
  METHOD 2: No DC at 6 months-Not evaluable/missing | 20.2 | 20.0 | 22.2 | 20.6

8. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) at 12 months based on BICR assessments according to RECIST v1.1. DCR at 6 months was evaluated using 2 different approaches to the length of stable disease (SD). -Method 1: Patients who had a best objective response of complete response (CR) or partial response (PR) within 24 weeks or had demonstrated SD for a minimum interval of 24 weeks following randomization. -Method 2: Patients who had a best objective response of CR or PR in the first 24 weeks or who had demonstrated SD for a minimum interval of 16 weeks following randomization.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 129 | 65 | 63 | 257
% participants
  DC at 12 months | 10.1 | 12.3 | 1.6 | 8.6
  No DC at 12 months | 89.9 | 87.7 | 98.4 | 91.4
  No DC at 12 months-Not evaluable/missing | 20.2 | 20.0 | 22.2 | 20.6

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression status at 6 months based on BICR assessments according to RECIST v1.1 at time of Progression Free Survival (PFS) analysis. Progression was defined as the time from the data of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdrew from therapy or received another anti-cancer therapy prior to progression. -Target Lesions, Non Target Lesions and New Lesions are not necessarily mutually exclusive categories. -Progression death refers to death in the absence of RECIST 1.1 progression.
Time Frame: After 6 months
Population: Full analysis set - all randomized patients
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 133 | 67 | 67 | 267
% participants
  Progression-Total | 82.0 | 82.1 | 88.1 | 83.5
  Total-RECIST 1.1 Progression | 57.9 | 59.7 | 67.2 | 60.7
  RECIST 1.1 progression-Target Lesions | 43.6 | 43.3 | 55.2 | 46.4
  RECIST 1.1 progression-Non-target lesions | 21.1 | 26.9 | 32.8 | 25.5
  RECIST 1.1 progression-New lesions | 26.3 | 20.9 | 26.9 | 25.1
  Progression-Death | 24.1 | 22.4 | 20.9 | 22.8
  No progression-Total | 18.0 | 17.9 | 11.9 | 16.5
  No progression-PD free and still being followed | 14.3 | 13.4 | 4.5 | 11.6
  No progression-Censored on Study Day 1 | 1.5 | 0 | 0 | 0.7
  No progression-Withdrawn consent | 0.8 | 3.0 | 1.5 | 1.5
  No progression- Censored death | 1.5 | 1.5 | 3.0 | 1.9
  No progression- Discontinued study | 0 | 0 | 3.0 | 0.7

10. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression status at 12 months based on BICR assessments according to RECIST v1.1 at time of Progression Free Survival (PFS) analysis. Progression was defined as the time from the data of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdrew from therapy or received another anti-cancer therapy prior to progression. -Target Lesions, Non Target Lesions and New Lesions are not necessarily mutually exclusive categories. -Progression death refers to death in the absence of RECIST 1.1 progression.
Time Frame: After 12 months
Population: Full analysis set - all randomized patients
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 133 | 67 | 67 | 267
% participants
  Progression-Total | 88.7 | 83.6 | 89.6 | 87.6
  Total-RECIST 1.1 Progression | 64.7 | 59.7 | 68.7 | 64.4
  RECIST 1.1 progression-Target Lesions | 50.4 | 47.8 | 56.7 | 51.3
  RECIST 1.1 progression-Non-target lesions | 23.3 | 28.4 | 32.8 | 27.0
  RECIST 1.1 progression-New lesions | 27.1 | 23.9 | 23.9 | 25.5
  Progression-Death | 24.1 | 23.9 | 20.9 | 23.2
  No progression-Total | 11.3 | 16.4 | 10.4 | 12.4
  No progression-PD free and still being followed | 6.8 | 11.9 | 3.0 | 7.1
  No progression-Censored death | 3.8 | 0 | 3.0 | 2.6
  No progression-Withdrawn consent | 0.8 | 4.5 | 1.5 | 1.9
  No progression-Discontinued study | 0 | 0 | 3.0 | 0.7

11. Secondary Outcome: Overall Survival
Description: Survival status at time of overall survival analysis. 'Still in survival follow-up' includes patients known to be alive at data cut-off. 'Terminated prior to death' includes patients with unknown survival status or patients who were lost to follow-up.
Time Frame: After 12 months
Population: Full analysis set - all randomized patients
Measure: Number; unit: % participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 133 | 67 | 67 | 267
% participants
  Death | 64.7 | 65.7 | 76.1 | 67.8
  Still in survival follow-up | 30.1 | 28.4 | 16.4 | 26.2
  Terminated prior to death | 5.3 | 6.0 | 7.5 | 6.0
  Terminated prior to death-Voluntary discon. | 5.3 | 6.0 | 4.5 | 5.2
  Terminated prior to death-Other | 0 | 0 | 3.0 | 0.7

12. Secondary Outcome: Quality of Life
Description: Improvement in quality of life was assessed using European Organisation for Research and Treatment of Cancer (EORTC) questionnaires: -The impact of treatment on Health-Related Quality of Life, functioning, and symptoms was evaluated using the EORTC QLQ-C30 v3. -Head and neck cancer-specific symptoms were evaluated using the EORTC QLQ-H&N35. The symptom and QoL/function improvement rate was defined as the number (%) of patients with 2 consecutive assessments at least 14 days apart that showed a clinically meaningful improvement (a decrease from baseline score ≥10 or EORTC QLQ-C30 scales) in that symptom/function from baseline. For QLQ-H&N35A a minimum clinically meaningful change was defined as a change in the score from baseline of >10 for scales/items
Time Frame: After 12 months
Population: Full analysis set - all randomized patients
Measure: Number (95% Confidence Interval); unit: % patients
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab
Number analyzed (Participants) | 133 | 67 | 67
% patients
  EORTC QLQ-C30 Function-Physical | 12 [6.7 to 20.8] | 13.6 [6.4 to 26.7] | 5.1 [1.4 to 16.9]
  EORTC QLQ-C30 Function-Role | 16.3 [10.0 to 25.5] | 16.7 [8.3 to 30.6] | 11.8 [4.7 to 26.6]
  EORTC QLQ-C30 Function-Cognitive | 25 [16.2 to 36.4] | 29.4 [16.8 to 46.2] | 10.7 [3.7 to 27.2]
  EORTC QLQ-C30 Function-Emotional | 13.5 [7.9 to 22.1] | 13.6 [6.4 to 26.7] | 2.6 [0.5 to 13.2]
  EORTC QLQ-C30 Function-Social | 18.3 [11.0 to 28.8] | 15.2 [6.7 to 30.9] | 16.1 [7.1 to 32.6]
  EORTC QLQ-C30 Symptom-Fatigue | 16.8 [10.9 to 25.0] | 17.3 [9.4 to 29.7] | 7.5 [3.0 to 17.9]
  EORTC QLQ-C30 Symptom-Pain | 22.8 [15.4 to 32.4] | 20.8 [11.7 to 34.3] | 6.7 [2.3 to 17.9]
  EORTC QLQ-C30 Symptom-Nausea/vomiting | 22.2 [12.5 to 36.3] | 16.7 [4.7 to 44.8] | 17.6 [6.2 to 41.0]
  EORTC QLQ-C30 Global health status/QoL | 13.4 [8.3 to 20.9] | 7.3 [2.9 to 17.3] | 3.7 [1.0 to 12.5]
  EORTC QLQ-H&N35 Scale-Pain | 16.7 [9.8 to 26.9] | 19.4 [9.8 to 35.0] | 8.3 [2.9 to 21.8]
  EORTC QLQ-H&N35 Scale-Swallowing | 16.0 [9.4 to 25.9] | 13.3 [6.3 to 26.2] | 10.3 [4.1 to 23.6]
  EORTC QLQ-H&N35 Scale-Senses | 17.8 [10.7 to 28.1] | 24.3 [13.4 to 40.1] | 23.1 [12.6 to 38.3]
  EORTC QLQ-H&N35 Scale-Speech | 20.2 [13.3 to 29.4] | 9.8 [4.3 to 21.0] | 19.6 [10.7 to 33.2]
  EORTC QLQ-H&N35 Scale-Social eating | 21.3 [13.7 to 31.4] | 20.0 [10.9 to 33.8] | 15.0 [7.1 to 29.1]
  EORTC QLQ-H&N35 Scale-Social contact | 22.6 [14.0 to 34.4] | 5.9 [1.6 to 19.1] | 13.0 [4.5 to 32.1]
  EORTC QLQ-H&N35 Scale-Sexuality | 16.2 [9.5 to 26.2] | 9.5 [3.8 to 22.1] | 9.5 [3.8 to 22.1]

13. Secondary Outcome: Duration of Response
Description: Duration of objective response in patients with objective response based on BICR assessments according to RECIST v1.1. Duration of response was the time from the first documentation of Complete response/Partial response (which was subsequently confirmed) until the date of progression, death, or the last evaluable RECIST assessment for patients that did not progress. An ongoing response was defined as a patient who had documented objective response and was still alive and progression-free at the time of the data cut-off (per RECIST v1.1 as assessed by BICR).
Time Frame: After 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MEDI4736 + Tremelimumab | MEDI4736 | Tremelimumab | Total
Number analyzed (Participants) | 10 | 6 | 1 | 17
Participants
  No. progressed or died within 12 months | 5 | 2 | 0 | 7
  No. progressed or died after 12 months | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from time the informed consent was signed through 90 days after the last dose of the last study treatment or until another therapy was initiated.
Description: AEs were either spontaneously reported by the patient or reported in response to open questions, revealed by observation, or were changes from baseline/deterioration in tests and vital signs that met SAE criteria or led to IP discontinuation. AEs/SAEs were followed up for resolution after discontinuation or study completion and for as long as medically indicated. AE and SAE data are reported using the Safety Analysis Set.
Arm/Group | MEDI4736 AND TREMELIMUMAB COMBINATION | MEDI4736 | Tremelimumab
All-Cause Mortality (participants affected / at risk) | 86/133 | 44/67 | 51/67
Serious Adverse Events (participants affected / at risk) | 59/133 | 18/65 | 25/65
Other Adverse Events (participants affected / at risk) | 110/133 | 52/65 | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 AND TREMELIMUMAB COMBINATION (N=133) | MEDI4736 (N=65) | Tremelimumab (N=65)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocytic hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 0 (0) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 9 (10) | 1 (1) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exsanguination (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 AND TREMELIMUMAB COMBINATION (N=133) | MEDI4736 (N=65) | Tremelimumab (N=65)
Anaemia (Blood and lymphatic system disorders) | 20 (20) | 11 (14) | 11 (12)
Tachycardia (Cardiac disorders) | 5 (5) | 0 (0) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 4 (4)
Hypothyroidism (Endocrine disorders) | 15 (15) | 9 (9) | 6 (6)
Constipation (Gastrointestinal disorders) | 18 (19) | 9 (9) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 27 (42) | 12 (14) | 14 (19)
Dysphagia (Gastrointestinal disorders) | 14 (15) | 8 (9) | 6 (7)
Nausea (Gastrointestinal disorders) | 18 (24) | 7 (8) | 18 (22)
Vomiting (Gastrointestinal disorders) | 9 (13) | 4 (4) | 9 (11)
Asthenia (General disorders) | 21 (24) | 10 (12) | 8 (11)
Fatigue (General disorders) | 25 (29) | 19 (23) | 12 (12)
Mucosal inflammation (General disorders) | 1 (1) | 4 (4) | 1 (2)
Oedema peripheral (General disorders) | 7 (7) | 2 (3) | 2 (2)
Pain (General disorders) | 5 (5) | 0 (0) | 8 (8)
Pyrexia (General disorders) | 16 (19) | 5 (5) | 12 (16)
Weight decreased (Investigations) | 18 (18) | 5 (5) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 25 (27) | 10 (11) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 6 (10) | 0 (0) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (8) | 6 (7) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (10) | 3 (3) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (6) | 5 (5) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 4 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (4) | 6 (8)
Dizziness (Nervous system disorders) | 4 (5) | 3 (3) | 5 (6)
Headache (Nervous system disorders) | 6 (7) | 6 (7) | 7 (7)
Paraesthesia (Nervous system disorders) | 3 (3) | 5 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9) | 3 (3) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (10) | 12 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (15) | 6 (6) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 3 (3) | 5 (6)
Hypertension (Vascular disorders) | 8 (11) | 6 (7) | 1 (1)
Hypotension (Vascular disorders) | 7 (7) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publications prior to public release for a period up to 120 days to confirm accuracy, prevent disclosure of confidential information, and ensure that information is handled appropriately.